CLINICAL TRIAL: NCT06473688
Title: The DEXTER-assisted Non-emergent and Acute Cholecystectomy Study
Brief Title: The DEXTER-assisted Non-Emergent and Acute cholecyStecTomy Study (The NEST Study)
Acronym: NEST
Status: Completed | Type: Observational
Sponsor: Distalmotion SA (Industry)
Collaborators: Confinis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-02
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cholecystectomy
MeSH Terms: interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cholecystectomy — Robotic-assisted and laparoscopic cholecystectomy

SUMMARY:
This study aims to confirm the perioperative and early postoperative safety and clinical performance (efficacy) of the Dexter Robotic System, in patients undergoing robotic-assisted and laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Patients planned to undergo elective robot-assisted and laparoscopic cholecystectomy; using one camera port, two ports for the manipulating instruments, and additional ports as needed.

Exclusion Criteria:

* Morbidly obese patients (BMI > 40)
* Any relative and absolute contraindications for the use of conventional endoscopes and endoscopic surgical instruments
* Need for robotic stapling, advanced energy delivery, ultrasound, cryoablation and microwave energy delivery
* Bleeding diathesis
* Pregnancy
* Patients with pacemakers or internal defibrillators
* Any planned concomitant procedures
* Patient deprived of liberty by administrative or judicial decision
* Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing a cholecystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
primary safety endpoint | up to 30 days
  occurrence of Clavien - Dindo grades III-V adverse events
primary performance endpoint | intraoperative
  successful completion of the Dexter-assisted procedure, i.e. free of any conversion to an open or fully laparoscopic surgical approach

CONTACTS AND LOCATIONS:
Locations (4):
- Groupe Hospitalier Saintes - Saint-Jean-d'Angély, Saintes, France
- Universitätsklinikum Bonn, Bonn, Germany
- Switzerland (2):
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No